CLINICAL TRIAL: NCT02230462
Title: Effects of Visualization of Pre-operative Defects on Patient Satisfaction After Facial Reconstruction for Skin Cancer Resection.
Brief Title: Patient Satisfaction After Facial Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H13-02922
Record Dates: First submitted 2014-07-16; First posted 2014-09-03 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Skin Neoplasms
Keywords: patient satisfaction; Mohs surgery
MeSH Terms: conditions — Skin Neoplasms; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viewing of cancer excision defect (Experimental): Patients in this arm of the study will be invited to view their cancer excision defect, with the aid of a mirror, prior to its reconstruction.
  Interventions: Other: Viewing of cancer excision defect
- No viewing of cancer excision defect (No Intervention): Patients in this arm of the study will not be invited to view their cancer excision defect prior to its reconstruction.

INTERVENTIONS:
Other: Viewing of cancer excision defect — Patients will be invited to view their cancer excision defect, with the aid of a mirror, prior to its reconstruction.
  Arms: Viewing of cancer excision defect

SUMMARY:
The purpose of this study is to assess the effects of visualization of skin cancer resection defects on the face on the post-operative satisfaction of patients after their reconstruction. To achieve this aim, patients invited to participate in this study will be randomized to either seeing or not seeing their skin cancer excision defect prior to reconstruction. After reconstruction, patient satisfaction will be assessed in both groups to determine if visualization of the defect prior to reconstruction has any effect on patient satisfaction and if any detected effect has durability over time.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to assess patient satisfaction after reconstruction of Mohs skin cancer resection defects in the face, with the resection defect either seen or unseen by the patient. In this way, the investigators will determine the effects of visualization of the pre-operative defects on patient satisfaction after facial reconstruction. Any effects on patient satisfaction that are identified will then be tracked over time.

Hypothesis:

The null hypothesis for this study is that patient satisfaction after reconstruction of Mohs defects on the face is unaffected by the opportunity to visualize the defect prior to reconstruction, and that this observation persists over time. Furthermore, patients are able to recall the size of their cancer resection defect as accurately from a detailed description as from seeing the defect in a mirror.

Justification:

This study will address whether visualization of a defect prior to its reconstruction affects patient satisfaction. Visualization of a defect prior to reconstruction is not standardized and is occasionally, but by no means necessarily, a portion of their consent for the reconstruction procedure. For the excision and reconstruction procedure in this study, all patients will be receiving the gold standard treatment for skin cancer. This includes a Mohs excision of their cancer and subsequent reconstruction of the excision defect using either primary closure or local flaps. Alternative treatments to this approach include various forms of excision and reconstruction where cancer free margins cannot be immediately determined.

Objectives:

The objectives of this study are to determine whether visualization of a cancer excision defect on the face, prior to its reconstruction, improves post-reconstruction patient satisfaction. The satisfaction measures sought will primarily be satisfaction with the cosmetic result but will also include measures pertaining to symptomatic scarring, skin related quality of life and ability to recall defect size will also be collected.

Research Method:

Patients meeting research criteria will be recruited to this study. These patients will all undergo cancer excision and reconstruction of the skin cancer defect during the same clinic visit. After their cancer excision is complete, they will be and randomized to either viewing or not-viewing their skin cancer excision defect prior to its reconstruction. After reconstruction they will be provided a series of surveys that assess the research questions posed by this study. Surveys will be distributed in the clinic on the day of surgery and at routine follow-up appointments at one week and two to three months.

Statistical Analysis:

The planned sample size for this study is eighty patients randomized to two groups of forty. Study end points will be sought from patient answers to three sets of surveys that determine patient satisfaction with the cosmetic appearance of their reconstruction, ranked on an ordinal scale, as a primary end-point. Secondary end points using ordinal and binary measures will also be sought and include skin related quality of life (as measured by the Skindex 16), scarring, and the ability to accurately recall the size of the skin cancer excision defect. A chi-squared analysis of the data will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients recruited for this study must undergo Mohs resection of skin cancer of the face with negative margins at the completion of their cancer resection.
* Patients recruited for this study must have a post cancer resection defect on the face at least 1.5 centimeters in size in the greatest dimension.
* Patients recruited for this study must undergo single stage repair of their post cancer resection defect with primary closure or local flaps.
* Patients must be from the Greater Vancouver area.

Exclusion Criteria:

* Patients with insufficient visual acuity to be able to appreciate wound and scarring changes to their face post-operatively will be excluded.
* Patients lacking the cognitive capacity to complete the data collection forms utilized in this study will be excluded.
* Patients suffering from significant psychiatric conditions will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with the cosmetic appearance of their skin cancer reconstruction. | The day of reconstruction.
  Patient satisfaction with the cosmetic appearance of their skin cancer reconstruction site will be assessed on a ten point scale on the day of surgery.

SECONDARY OUTCOMES:
Ability to recall cancer excision defect size. | 3 months after reconstruction
  Patients will be asked to draw what they recall to be the size of their cancer excision defect prior to its reconstruction. This will be done at the final routine surgical follow up appointment (3 months after surgery).
Symptomatic scarring | 3 months after reconstruction
  Patients will complete survey questions to determine whether they are bothered by their scar appearance, texture or any neuropathic symptoms.
Persistence of patient satisfaction with the cosmetic appearance of their skin cancer reconstruction. | 2 weeks, and 3 months after reconstruction.
  Patient satisfaction with the cosmetic appearance of their skin cancer reconstruction site will be reassessed on a ten point scale at the two week and 3 month routine followup appointments.

OTHER OUTCOMES:
Skindex -16 | The day of reconstruction, 2 weeks, and 3 months after reconstruction.
  Patient quality of life relating to their skin cancer will be assessed using the Skindex-16 (a validated tool for this purpose).

CONTACTS AND LOCATIONS:
Overall Officials: Bryce J Cowan, MD, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Dermatology & Skin Science (UBC), The Skin Care Centre, Vancouver, British Columbia, Canada